CLINICAL TRIAL: NCT00708656
Title: A Randomized, Single-Blind Study to Assess Efficacy and Safety of Dosing Mesalazine 800 mg Tablets (Asacol®) at 2.4 g Once Daily Versus Divided Doses 3 Times Daily for 12 Months in Maintenance of Remission of Ulcerative Colitis.
Brief Title: The Colitis Once Daily Asacol Study
Acronym: CODA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAW0105; ISRCTN:35600632; EudraCT Number:2005-002784-91
Record Dates: First submitted 2008-04-08; First posted 2008-07-02 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2010-09

CONDITIONS: Ulcerative Colitis
Keywords: IBD; Colitis; UC
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: once daily (Experimental): Three 800mg tablets of mesalazine (Asacol®) in the morning
  Interventions: Drug: mesalazine (Asacol®)
- 2: tds (Active Comparator): Mesalazine (Asacol®) 800mg given three times daily
  Interventions: Drug: mesalazine (Asacol®)

INTERVENTIONS:
Drug: mesalazine (Asacol®) — 800 mg tablets
  Other Names: Mesalazine; Asacol

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of dosing mesalazine 800 mg tablets (Asacol®) at 2.4 g once daily versus divided doses three times daily in the maintenance of remission of ulcerative colitis.

DETAILED DESCRIPTION:
Study design

* Multicentre, randomized, single-blind, comparator-controlled, parallel-armed study
* One year follow-up, or until relapse (whichever shorter)
* 40-60 UK centres

Subject population

* Ulcerative colitis in remission (sigmoidoscopy score of 0 or 1 with no symptoms of active disease, with no treatment for active colitis) for at least 4 weeks, and for no more than 2 years
* Taking mesalazine or sulfasalazine prior to study entry
* Patients excluded if they have Crohn's disease, symptoms of active colitis, have used corticosteroids, ciclosporin or oral/enema mesalazine in the past 4 weeks, are intolerant to mesalazine or Asacol, are pregnant or lactating, or have known HIV, hepatic disease, renal impairment or other serious medical or psychiatric illness
* Sample size 250
* Gender: male or female
* Ethnicity: no restriction
* Age: over 18

Test Product

Once daily group: Asacol® 2.4g daily given as three 800mg tablets orally qAM

Three times daily group: Asacol® 2.4g daily given as one 800mg tablet orally three times daily

Criteria for Evaluation:

Primary Outcome Variable: Relapse rate over 1 year in the intention to treat population, with the study powered to detect non-inferiority of the once-daily regimen.

Secondary Outcome Variables: assessment of superiority of the once-daily regimen, if non-inferiority is demonstrated; safety analysis; per protocol analysis of relapse rate; time course of relapse; medication compliance; changes in modified Baron sigmoidoscopy scores between trial entry and relapse/12 month; impact of various factors on relapse rate (time from last relapse at study entry, concomitant azathioprine or 6-mercaptopurine therapy; disease extent; disease duration; smoking status; age at diagnosis; previous dose of mesalazine; baseline calprotectin; baseline CRP level).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria will be eligible for study entry:

* Male and female patients aged over 18 with ulcerative colitis confirmed by histology who are in remission (no symptoms of active disease, and modified Baron sigmoidoscopic score of 0 or 1)
* If female, must be (as documented in patient notes):

  * postmenopausal (at least 1 year without spontaneous menses), or
  * surgically sterile (tubal ligation or hysterectomy at least 6 months prior to enrollment), or
  * using acceptable contraception (e.g., oral, intramuscular, or implanted hormonal contraception) at least 3 months prior to enrollment, or
  * have a sexual partner with non-reversed vasectomy (with confirmed azoospermia), or
  * be using 1 barrier method (e.g., condom, diaphragm, spermicide, or intra-uterine device)
* Patients whose ulcerative colitis has been in clinical remission for 4 weeks or longer, and who have had a symptomatic relapse within the past two years
* Patients taking mesalazine, sulfasalazine or other drug containing 5-ASA for 4 weeks or longer
* Patients capable of giving written informed consent

Exclusion Criteria:

The following patients will be excluded from the study:

* Patients with Crohn's disease
* Patients with symptoms of active colitis
* Modified Baron sigmoidoscopy score of 2 or 3
* Patients who have used oral, enema, intravenous or suppository preparations of corticosteroids, oral or intravenous ciclosporin, mesalazine enemas or suppositories within the past four weeks
* Patients taking azathioprine or 6-mercaptopurine who have altered the dose or started treatment within the past three months, (these drugs permitted in stable dose during the study)
* Patients with intolerance to Asacol 400 mg or mesalazine
* Women who are pregnant or lactating
* Patients with known HIV infection
* Patients with hepatic disease
* Patients with renal impairment (creatinine above local reference range), or with positive urine dipstick test to blood or protein
* Other serious medical or psychiatric illness that in the opinion of the investigator would possibly comprise the study
* Patients with problem alcohol excess or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2006-10; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To assess whether a once daily dose of three 800mg tablets of mesalazine (Asacol®) in the morning is equivalent to mesalazine (Asacol®) given as 800mg three times daily in preventing relapse over a 12 month period. | At relapse or 12 month follow up

SECONDARY OUTCOMES:
To assess equivalence in terms of safety | 12 months
To assess equivalence in terms of time to relapse | 12 months
To assess equivalence in terms of progression of disease (measured by Mayo score) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr A B Hawthorne, Principal Investigator — Cardiff and Vale University Health Board; Professor C Probert, Principal Investigator — Bristol Royal Infirmary
Locations (45):
- United Kingdom (45):
  - Barnsley District General Hospital, Barnsley
  - North Hampshire Hospital, Basingstoke
  - Birmingham Heartlands Hospital, Birmingham
  - Selly Oak Hospital, Birmingham
  - Bishop Auckland General Hospital, Bishop Auckland
  - Blackpool Victoria Hospital, Blackpool
  - Glan Clwyd Hospital, Bodelwyddan
  - Pilgrim Hospital, Boston
  - Princess Royal Hospital, Brighton
  - Royal Sussex County Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - Llandough Hospital, Cardiff
  - University Hospital of Wales, Cardiff
  - Cumberland Infirmary, Carlisle
  - Walsgrave Hospital, Coventry
  - Derby City General Hospital, Derby
  - Dr M Al-Najjar, Doncaster
  - Russells Hall Hospital, Dudley
  - University Hospital of North Durham, Durham
  - Stobhill Hospital, Glasgow
  - Gloucester Royal Hospital, Gloucester
  - University Hospital of Hartlepool, Hartlepool
  - Hull Royal Infirmary, Hull
  - Royal Glamorgan Hospital, Llantrisant
  - County Hospital, Louth
  - Luton & Dunstable Hospital, Luton
  - Macclesfield District General Hospital, Macclesfield
  - Borders General Hospital, Melrose
  - Prince Charles Hospital, Merthyr Tydfil
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Derriford Hospital, Plymouth
  - Poole General Hospital, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Rotherham District General Hospital, Rotherham
  - Royal Hallamshire Hospital, Sheffield
  - University Hospital of North Tees & University Hospital of Hartlepool, Stockton-on-Tees
  - Royal Cornwall Hospital, Truro
  - Queen Elizabeth II Hospital, Welwyn Garden City
  - New Cross Hospital, Wolverhampton
  - Alexandra Hospital, Worcester
  - Worcester Royal Infirmary, Worcester
  - Worthing Hospital, Worthing
  - Yeovil District Hospital, Yeovil
  - York District Hospital, York

REFERENCES:
- [Derived] Gillespie D, Farewell D, Barrett-Lee P, Casbard A, Hawthorne AB, Hurt C, Murray N, Probert C, Stenson R, Hood K. The use of randomisation-based efficacy estimators in non-inferiority trials. Trials. 2017 Mar 9;18(1):117. doi: 10.1186/s13063-017-1837-3. PMID 28274254